CLINICAL TRIAL: NCT06510777
Title: A Pragmatic, Multi-centre, Prospective, Randomized, Superiority Study to Compare the Performance of the Single-use Negative Pressure Wound Therapy System PICO Versus Standard of Care in the Management of Venous Leg Ulcers
Brief Title: PICO Venous Leg Ulcers (VLU) Reimbursement Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Early terminated due to protocol design issues with inability to correct at this stage.
Sponsor: Smith & Nephew, Inc. (Industry)
Collaborators: CEN Biotech (Industry); T.J. Smith and Nephew, Limited (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PICO.2021.09; 2023-A01760-45 (Other: ANSM)
Record Dates: First submitted 2024-07-15; First posted 2024-07-19 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Venous Insufficiency; Venous Leg Ulcer
Keywords: Venous Leg Ulcer; Negative Pressure Wound Therapy; NPW; Hard-to-Heal Venous Leg Ulcer; Community Care
MeSH Terms: conditions — Venous Insufficiency; Varicose Ulcer | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The primary endpoint (i.e., 100% epithelialization) includes a blind assessment to reduce bias. The Blind Assessment Board will assess the primary endpoint using subject-series of wound photos, being unaware of treatment allocation of subjects.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PICO Treatment Arm (Experimental): The maximum duration for treatment with PICO will be 12 weeks.
  PICO treatment will be discontinued if the wound does not respond to treatment after 2 weeks according to predefined criteria, if the wound gets worse at any time, if the wound is 100% epithelialized, or if the wound presents advanced healing, which will be assessed using predefined criteria. In the latter case where the VLU is determined sufficiently healed according to the pre-specified criteria in the protocol, subjects will be switched to Standard of Care (SOC).
  Wound care treatment at home will be done by home care nurses. Compression therapy will be maintained throughout the entire patient's follow-up.
  Interventions: Device: PICO Treatment; Device: Standard of Care (SOC) Treatment
- Standard of Care Treatment Arm (Active Comparator): Wounds are treated with appropriate traditional dressings throughout the study based on wound condition and healing trajectory. Wound care treatment at home will be done by home care nurses. Compression therapy will be maintained throughout the entire patient's follow-up.
  Interventions: Device: Standard of Care (SOC) Treatment

INTERVENTIONS:
Device: PICO Treatment — PICO 7 is a single-use Negative Pressure Wound Therapy System consisting of a small portable pump, 2 AA batteries, 1 or 2 dressings, and fixation strips. The dressing is changed when the dressing is saturated or after 7 days of treatment.
  PICO Treatment will be given in addition to compression therapy.
  If the wound is healed and until the wound healing confirmation visit, Venous Leg Ulcers (VLUs) allocated to the PICO group may be covered using a protective dressing.
  If the wound meets the wound improvement criteria as assessed by the PI during the monthly visits, PICO treatment may be stopped.
  Other Names: Single-Use Negative Pressure Therapy System PICO 7 (sNPWT)
  Arms: PICO Treatment Arm
Device: Standard of Care (SOC) Treatment — Application of an appropriate wound primary dressing according to its intended purpose and chosen appropriately according to wound healing stage:
  1. Dressing choice should take wound condition into consideration but may also consider subject's comfort (including pain) and HCP's preference.
  2. Sequential treatment:
     * Debridement stage: alginate, hydrogel, absorbent, or hydro-detersive dressings
     * Granulation stage: wound contact layer, foam, petrolatum, or hydrofiber dressings
     * Epithelialization stage: wound contact layer, hydrocolloids
     * Other: dressings for specific clinical situations (e.g. fragile skin, infection; hemorrhagic wound, malodorous wound)
  3. Application of appropriate venous compression therapy based on Ankle Brachial Pressure Index (ABPI) value.
  Other Names: Traditional wound dressings in addition to compression therapy.

SUMMARY:
This study intends to demonstrate the superiority of PICO treatment when applied up to 12 weeks, versus Standard of Care (SOC) in the treatment of hard to heal Venous Leg Ulcers (VLU) by community-based practitioners. The primary endpoint is the incidence of confirmed healed VLUs at 12 weeks or before, in the PICO treatment group versus the SOC group. The study hypothesis is based on the Kirsner study (Kirsner R, Dove C, Reyzelman A, Vayser D, Jaimes H. A prospective, randomized, controlled clinical trial on the efficacy of a single-use negative pressure wound therapy system, compared to traditional negative pressure wound therapy in the treatment of chronic ulcers of the lower extremities. Wound Repair Regen. 2019 Sep;27(5):519-529)), which compared PICO treatment to traditional NPWT (t-NPWT); the ITT analysis in the subgroup of patients with VLU showed 45.1% wound closure (confirmed wound healing) at 12 weeks in the PICO group as compared to 28% in the t-NPWT group, yielding a difference of 17.1%, 95% Confidence Interval = (-1.9%;+35.4%). For our study, the Sponsor made the assumptions that the t-NPWT healing proportion (28%) can be used as conservative estimate for the control group proportion and that the PICO group should provide at least a 17% improvement over standard of care. Adaptative design is chosen to adjust the sample size using the re-assessment size method to preserve alpha risk (α) level.

DETAILED DESCRIPTION:
This is a national, multicentre, pragmatic, randomized, controlled superiority study in which PICO treatment with compression therapy will be compared against Standard of Care (i.e. traditional wound dressings with compression therapy). There will be two parallel treatment arms with a 1:1 allocation ratio and a stratification on wound duration and size. There will be an additional blind assessment for the primary outcome measure.

Approximately 37 investigational sites located in France will be enrolled. At each site, a community-based practitioner (general practitioner or specialist) will be enrolled as Principal Investigator (PI). District nurses will be responsible for providing wound care in homecare setting. Duly informed and eligible patients will complete an inclusion visit after which they will enter in a 2-week run-in period in which subjects will be treated with standard of care. After these 2 weeks of run-in, eligibility to randomization will be assessed using pre-specified criteria listed in the protocol, that aim to confirm that the wound does not respond to an adequately conducted standard of care in a satisfactory manner, including subject compliance with compression therapy.

Upon randomization, baseline data will be collected, and each subject will be followed-up by the PI for 12 weeks. The PI will conduct 3 visits, i.e., at Week 4 (D28±3 days), Week 8 (D56±3 days), and Week 12 (D84±3 days). Relevant study data will be collected at these visits. In the event wound healing is observed during the 12-week follow-up period of the study either by the PI or by the home care nurse, a Wound Healing Confirmation Visit needs to be conducted with the PI 2 weeks later (±3 days) to confirm that the wound is still healed. Only wounds still healed at the wound healing confirmation visit will be counted as "healed" in the primary endpoint analysis. This means that for wounds that are not healed by Week 12, the visit with the PI at Week 12 will be the final study visit for the subject. Following, because a Wound Healing Confirmation Visit needs to be conducted 2 weeks (±3 days) following the initial observation of wound healing, which can occur at any time throughout the 12 week follow-up period, the Wound Healing Confirmation Visit can occur at any time as well, but at the latest 2 weeks (±3 days) following the visit at Week 12, i.e. at week 14±3 days.

In between study visits with the PI, patients are cared for at home by their home care nurse who will also be trained on the study. The study nurse will be collecting study related data as well using a secure mobile application.

ELIGIBILITY:
Inclusion Criteria:

* Subject signed informed consent
* Both gender adult ≥ 18 years old
* Venous leg ulcer (VLU) diagnosed by:

  * ABPI ≥ 0.7 and < 1.3 within the last 3 months
  * If ABPI < 1.3, one of the following measures should be available:

    * Toe Brachial Pressure Index (TBPI) > 0.7
    * Toe pressure (TP) > 50 mmHg
    * Transcutaneous oxygen pressure (TcPO2) > 30 mmHg
* VLU duration ≥ 6 weeks
* VLU surface area:

  * Isolated leg ulcer: ≤ 100 cm^2
  * Non-isolated leg ulcers: pooled surface area ≤ 100 cm^2 that can be covered by a single dressing
* Exuding VLU according to clinical judgement
* The subject is in acceptable state of health and nutrition according to clinical judgement
* The subject is able to follow the protocol instruction and willing to comply with compression therapy
* The subject is affiliated to a French Health insurance scheme

Exclusion Criteria:

* Clinical evidence of VLU infection [i.e. presence of at least 3 overt signs of local infection (e.g., erythema, warmth, swelling, pain, odor) or signs of spreading or systemic infection)
* Wound with necrotic tissue after debridement
* Sloughy wound (100% of slough) after debridement
* Exposed arteries, veins, nerves or organs
* Current therapy with chronic oral corticosteroids (>10 days)
* Previous therapy with negative pressure wound therapy device or hyperbaric oxygen within 7 days prior to enrolment
* Arterial insufficiency non-revascularized
* Wound actively bleeding
* Malignant wound
* Enrolled in another clinical trial or being in a period of exclusion from a previous clinical trial
* Person belonging to a population referred to in articles 64 (incapacitated subjects), 65 (minors), 66 (pregnant or breastfeeding women), 67 (persons performing mandatory military service, persons deprived of liberty, persons who, due to a judicial decision cannot take part in clinical investigations) and 68 (patients in emergency situation) of the Medical Device Regulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 142 (Actual)
Dates: Start 2023-12-29 (Actual); Primary Completion 2025-10-24 (Actual); Study Completion 2025-10-24 (Actual)

PRIMARY OUTCOMES:
Number of Venous Leg Ulcers (VLUs) confirmed healed by or at 12 weeks | Up to 12 weeks
  The primary endpoint is the incidence of confirmed healed Venous Leg Ulcers (VLUs) at 12 weeks or before in PICO versus SOC group.
  A confirmed healed VLU is defined as a wound with complete closure (100% epithelialization) according to PI's judgement during two visits that are two weeks apart (±3 days) AND confirmed by a blind assessment board based on blinded photograph examination.

SECONDARY OUTCOMES:
Time to Achieve Wound Healing | Up to 12 Weeks
  Number of days required from baseline to achieve wound healing where the wound is observed with complete closure (100% epithelialization).
Relative Wound Area Reduction (RWAR) | Day 0, Week 4, Week 8, Week 12 (up to 14 weeks ±3days)
  Relative wound area reduction (RWAR) at Week 4, Week 8 and at the Final Visit i.e., visit at Week 12 or the Wound Healing Confirmation Visit.
Time to achieve 100% healthy granulation tissue | Day 0, Week 4, Week 8, Week 12 (up to 14 weeks ±3 days)
  Number of days required to achieve 100% granulation over 12 weeks
Changes in quality of life using the generic EuroQol 5 Dimension (EQ-5D-5L ) | Day 0 to Week 12 (up to 14 weeks ±3 days)
  Changes in quality of life from baseline to the final visit (i.e., the visit at Week 12 or the Wound Healing Confirmation Visit).
  The descriptive system is used to describe the subject's health state & consists of 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels to choose the most appropriate answer: no problems, slight problems, moderate problems, severe problems, and extreme problems. The subject is asked to indicate his/her health state by marking the most appropriate statement in each of the five areas. Responses are coded as single-digit numbers expressing the severity level selected in each dimension. For instance, 'slight problems' (e.g. 'I have slight problems in walking about') is always coded as '2'. The digits for the 5 dimensions are combined in a 5-digit code. A higher number is a better outcome.
Changes in quality of life using the disease specific VEINES-Qol (Venous Insufficiency Epidemiological and Economic Study on Quality of Life) questionnaire | Day 0 to Week 12 (up to 14 weeks ±3 days)
  Changes in quality of life from baseline to the Final Visit (i.e., the visit at Week 12 or the Wound Healing Confirmation Visit).
  The VEINES-QOL questionnaire consists of 26 items. It includes questions about symptoms due to Chronic Venous Disorders of the Leg (CVDL) (ten items), limitations in daily activities due to CVDL (nine items) and psychological impact (five items), as well as questions asking about the amount of change in the respondent's leg problem over a 1-year period (one item) and the time of day that the leg problem is most intense (one item).
  Of the 26 items in the questionnaire, 25 items are combined to create a summary score (VEINES-QOL). One item which asks about the time of day the leg problem is most intense (question 2), provides only descriptive information and is not scored. High values indicate better outcomes.
Number of Adverse Events | Day 0 to Week 12 (up to 14 weeks ±3 days)
  Number of participants with an adverse event
Number of device deficiencies | Day 0 to Week 12 (up to 14 weeks ±3 days)
  Number of participants with a device deficiency
Visual Analog Scale (VAS) score at dressing removal (PICO Treatment Arm only) | Day 0 to Week 12 (up to 14 weeks±3 days)
  Pain scores on removal of the dressing measured using a 0-100 Visual Analog Scale (VAS) score, with zero (0) indicating no pain and 100 indicating the worst possible pain.
VLU treatment impact on mobility and physical activity using a 5 point-Likert scale | Week 4, Week 8, Week 12 (up to 14 weeks±3 days)
  Venous Leg Ulcers (VLU) treatment impact on mobility and physical activity using a 5 point-Likert scale: (1) Strongly disagree, (2) Disagree, (3) Neither agree nor disagree, (4) Agree, or (5) Strongly agree)
Healthcare Practitioner (HCP) satisfaction assessed using a 5 point-Likert scale questionnaire | Week 12 (up to 14 weeks±3 days)
  Analysis of HCP satisfaction with PICO treatment assessed using a 5 point-Likert scale questionnaire (PICO treatment group only): (1) Strongly disagree, (2) Disagree, (3) Neither agree nor disagree, (4) Agree, or (5) Strongly agree)
Subject satisfaction assessed using a 5 point-Likert scale questionnaire | Week 12 (up to 14 weeks ±3 days)
  Analysis of subject satisfaction with PICO treatment assessed using a 5 point-Likert scale questionnaire (PICO treatment group only): (1) Strongly disagree, (2) Disagree, (3) Neither agree nor disagree, (4) Agree, or (5) Strongly agree)

OTHER OUTCOMES:
Cost-Effectiveness Analysis of VLU-Treatment in Community Setting | Day 0 to Week 12 (up to 14 weeks ±3 days)
  Comparison of the direct costs estimated from treatment initiation day until the Final Visit (i.e. visit at Week 12 or the Wound Healing Confirmation Visit).

CONTACTS AND LOCATIONS:
Overall Officials: Fleur Derdeyn, Study Director — Smith & Nephew, Inc.
Locations (44):
- France (44):
  - Clinique de L'Atlantique, Puilboreau, France
  - Cabinet Médical, Vandœuvre-lès-Nancy, France
  - Synartis, Aire-sur-la-Lys
  - Polyclinique de Picardie, Amiens
  - Cabinet Privé, Antibes
  - Clinique d'Argonay, Argonay
  - Cabinet de Médecine Vasculaire - Angiologie, Arignac
  - Clinique Rhône Durance, Avignon
  - Cabinet Médical, Béziers
  - Cabinet de Médecine Vasculaire, Bourg-en-Bresse
  - Cabinet Médical, Cahors
  - GCS Pôle Santé de Cahors, Cahors
  - Cicadom, Challes-les-Eaux
  - Sui'vui Santé, Château-Renault
  - Cabinet Médical Gambetta Paymal (CMPG), Clichy
  - CICA+, Dardilly
  - Maison de Santé d'Etauliers, Étauliers
  - Cicadom, Guilherand-Granges
  - Cabinet Privé, Idron
  - Clinique St. Charles, La Roche-sur-Yon
  - Cabinet Médical, Langon
  - Cicadom, Le Coteau
  - Clinique des Augustines, Malestroit
  - Pôle Santé, Montélimar
  - Cabinet Médical, Paris
  - One Clinic, Plaisir
  - Cabinet d'angiologie de Pont-l'Abbé, Pont-l'Abbé
  - Cabinet privé, Pontcharra
  - Cabinet Privé, Rambouillet
  - Centre de Médecine Vasculaire, Rodez
  - Cabinet Médical, Saint-Alban
  - Clinique Megival, Saint-Aubin-sur-Scie
  - Clinique Mégival, Saint-Aubin-sur-Scie
  - Cabinet Privé, Saint-Gély-du-Fesc
  - Cicadom, Saint-Nazaire
  - Cabinet d'Angiologie et de Médecine Vasculaire, Saint-Priest
  - Polyclinique de Picardie, Sainte-Maxime
  - Cabinet Privé, Sarreguemines
  - Centre Privé de Consultations Médico-Chirurgicales, Saumur
  - Cabinet Privé Soyaux, Soyaux
  - Cabinet Médical, Thionville
  - Clinique Pasteur, Toulouse
  - Centre Léon Blum, Villeurbanne
  - Cabinet Médical, Wattignies

IPD SHARING:
Plan to Share IPD: No